CLINICAL TRIAL: NCT05892926
Title: A Multicenter Observational Retrospective Study of Therapeutic Approaches and Clinical Outcomes in Real Clinical Practice in Russian Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Locally Advanced/Metastatic Gastric and/or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: HER2-positive Locally Advanced/Metastatic Gastric and/or Gastroesophageal Junction (GEJ) Adenocarcinoma in Russia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00028
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter non-interventional observational retrospective study with secondary data collection

DETAILED DESCRIPTION:
It will be multicenter study. Planned number of study sites is about 50 oncological centers specialized on anticancer chemotherapy in various regions of Russia. A multi-center collaborative effort will help to describe characteristics of patients with HER2-positive gastric and/or GEJ adenocarcinoma in different regions in the most comprehensive way and to capture more patients into database, not only limited to a single institution

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced/metastatic gastric and/or gastroesophageal junction (GEJ) adenocarcinoma, with the diagnosis established between the 1st January 2022 and the 1st January 2023.
* Patients with documented HER2+ status based on IHC score ± ISH status.
* Patients have an adequate archival tumor sample and slides suitable for reassessment HER2 status by the reference laboratory.
* Age ≥ 18 years at the time of inclusion.
* Patients provided written consent allowing for data and samples to be used in the future and this study would be covered by the consent for future use in accordance with ICH GCP, GPP (Good Pharmacoepidemiology Practices) and local law prior to inclusion in the study. If the patient is deceased, a waiver may be accepted.

Exclusion Criteria:

* Patients receiving trastuzumab deruxtecan currently or in the anamnesis.
* The participation in any randomized controlled trial within period since diagnosis (between the 1st January 2022 and the 1st January 2023) until the timepoint of data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 adult patients with HER2-positive locally advanced/metastatic gastric and/or gastroesophageal junction cancer who are monitored and treated
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
To describe the clinical and demographic profiles of patients with HER2-positive locally advanced or metastatic gastric/GEJ adenocarcinoma in the Russian Federation | 6 months

SECONDARY OUTCOMES:
To describe data on the diagnostic algorithms and therapeutic tactics in patients with HER2-positive locally advanced or metastatic gastric/GEJ adenocarcinoma in routine practice in the Russian Federation | 6 months
To describe data on the treatment approach in patients with HER2-positive locally advanced or metastatic gastric/GEJ adenocarcinoma in routine practice in the Russian Federation | 6 months
To assess the treatment outcomes of patients with HER2-positive locally advanced or metastatic gastric/GEJ adenocarcinoma in routine practice in the Russian Federation | 6 months
To characterize the concordance between HER2 IHC scores & ISH in local and reference laboratories | 6 months

CONTACTS AND LOCATIONS:
Locations (31):
- Russia (31):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Belgorod
  - Research Site, Chelyabinsk
  - Research Site, Chita
  - Research Site, Grozny
  - Research Site, Irkutsk
  - Research Site, Kaluga
  - Research Site, Kemerovo
  - Research Site, Khabarovsk
  - Research Site, Khanty-Mansiysk
  - Research Site, Kostroma
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Maykop
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Omsk
  - Research Site, Perm
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Severodvinsk
  - Research Site, Sochi
  - Research Site, Surgut
  - Research Site, Tomsk
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Ulan-Ude
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yuzhno-Sakhalinsk

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HR00028&attachmentIdentifier=fb28dbeb-34e9-4131-8efe-9e7fd4b79c76&fileName=D133HR00028_Study_report_Synopsis_2025_06_20_1_1.pdf&versionIdentifier=